CLINICAL TRIAL: NCT00678743
Title: An Open-label Extension of a Randomized, Double-blind, Placebo-controlled, Crossover Study to Evaluate Simvastatin 20 mg Plus Omacor 4g Compared to Simvastatin 20 mg Plus Placebo in Subjects With Mixed Dyslipidemia
Brief Title: An Open-label Extension to Assess the Continued Efficacy of Omacor Plus Simvastatin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Provident Clinical Research (Other)
Collaborators: Reliant Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Kevin C. Maki, PhD, Study Director/Chief Science Officer, Provident Clinical Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRV-06009X
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Results first posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Dyslipidemias
Keywords: cholesterol; dyslipidemia; omega 3
MeSH Terms: conditions — Dyslipidemias | interventions — Omacor; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Omacor 4 grams/day plus simvastatin 80 mg/day. (Other): Subjects who had successfully completed a 12-wk double-blind crossover study of P-OM3 plus simvastatin 20 mg/d were eligible for the open-label extension study. Omacor 4 grams/day plus simvastatin 80 mg/day. Simvastatin dose adjusted at Investigator discretion after week 6.
  Interventions: Drug: Omacor + simvastatin

INTERVENTIONS:
Drug: Omacor + simvastatin — Omacor 4 grams/day plus simvastatin 80 mg/day. Simvastatin dose adjusted at Investigator discretion after week 6.
  Other Names: Omega-3-acid ethyl esters; Lovaza; Zocor

SUMMARY:
The primary objective of this trial is to assess the continued efficacy of Omacor co-administered with simvastatin for lowering non-high-density lipoprotein cholesterol (non-HCL-C) levels.

DETAILED DESCRIPTION:
The present trial is an open-label, uncontrolled extension to the previous trial (PRV-06009) which utilized a randomized,double-blind, two-period crossover design with eight clinic visits.

The current trial consists of nine clinic visits over 104 weeks. There will be two treatment periods in this study:

* Phase I: All subjects will receive simvastatin 80 md/d plus Omacor 4 g/d for the first six weeks of the trial.
* Phase II: All subjects will receive simvastatin (at a dose to be determined at the discretion of the Investigator) plus Omacor 4 g/d for the remainder of the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Must have met all relevant inclusion/exclusion criteria prior to and throughout the previous double-blind study (PRV-06009)
* Must have completed the previous double-blind study to week 12.
* Provide written informed consent and authorization for protected health information

Exclusion Criteria:

* Study drug compliance less than 50% in PRV-06009
* Any ongoing serious adverse event from PRV-06009

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-08; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C. Maki, PhD, Study Director — Provident Clinical Research

REFERENCES:
- [Derived] Maki KC, Lawless AL, Kelley KM, Dicklin MR, Kaden VN, Schild AL, Rains TM, Marshall JW. Effects of prescription omega-3-acid ethyl esters on fasting lipid profile in subjects with primary hypercholesterolemia. J Cardiovasc Pharmacol. 2011 Apr;57(4):489-94. doi: 10.1097/FJC.0b013e318210fca5. PMID 21297494

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-label P-OM3 + Simvastatin: All subjects received P-OM3 +simvastatin 80 mg/d through Week 6. Some subjects were assigned P-OM3 + simvastatin 80 mg/d after Week 6 at the discretion of the investigator.
Period: Phase I (First 6 Weeks)
Arm/Group | Open-label P-OM3 + Simvastatin
Started | 16 (17 subjects were enrolled but only 16 subjects received the treatment. One subject withdrew prior to receiving the treatment.)
Completed | 14
Not Completed | 2
Period: Phase II (Week 7 Through Week 104)
Arm/Group | Open-label P-OM3 + Simvastatin
Started | 14
40 mg/d Simvastatin (Some subjects were assigned P-OM3 + 40 mg/d simvastatin starting Week 7) | 7
80 mg/d Simvastatin (Some subjects maintained their regimen of P-OM3 + 40 mg/d simvastatin starting Week 7) | 7
Completed | 13
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Of the 17 participants who were eligible to enroll in the extension, 14 completed the initial six weeks of P-OM3 1 simvastatin 80 mg open-label extension and are included in the final analysis.
Arm/Group | Omacor 4 Grams/Day Plus Simvastatin 80 mg/Day.
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 30.4 (1.1)
Hypertension [Number; unit: participants] | 6
Type 2 Diabetes Mellitus [Number; unit: participants] | 4
High NCEP risk (non-HDL-C <130 mg/dL) [Number; unit: participants] | 5
Moderate NCEP risk (non-HDL-C <160 mg/dL) [Number; unit: participants] | 7
Low NCEP risk (non-HDL-C <190 mg/dL) [Number; unit: participants] | 2
Weight [Mean (Standard Deviation); unit: kg] | 81.4 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Median % Change in Non-HDL-C From Baseline to Week 6
Description: The primary efficacy endpoint will be the median percent change in non-HDL-C from baseline (average of weeks -2, -1, and 0) of the PRV-06009 (NCT00487591) double-blind study to Week 6 of PRV-06009X.
  Briefly, non-HDL-C was measured at Weeks -2, -1, and 0 from blood samples, and the concentrations of non-HDL-C in the blood at these timepoints were averaged to obtain baseline non-HDL-C concentration. Similarly, non-HDLC was measured at Week 6 from blood samples. Statistical analysis was performed comparing the change in non-HDL-C concentration from baseline to Week 6 and presented herein.
Time Frame: Week 6
Population: The results are from the 14 participants who were on Omacor 4 grams/day plus simvastatin 80 mg/day who completed Week 6.
Measure: Median (95% Confidence Interval); unit: Median percent change from baseline
Groups:
- Omacor 4 Grams/Day Plus Simvastatin 80 mg/Day.: Subjects who had successfully completed a 12-wk double-blind crossover study of P-OM3 plus simvastatin 20 mg/d were eligible for the open-label extension study. During the extension study, participants received Omacor 4 grams/day plus simvastatin 80 mg/day. Simvastatin dose adjusted at Investigator discretion after week 6 on Omacor 4 grams/day plus simvastatin 80 mg/day.
  Omacor + 80 mg/day simvastatin: Omacor 4 grams/day plus simvastatin 80 mg/day. Simvastatin dose adjusted at Investigator discretion after week 6 on Omacor 4 grams/day plus simvastatin 80 mg/day.
Arm/Group | Omacor 4 Grams/Day Plus Simvastatin 80 mg/Day.
Number analyzed (Participants) | 14
Median percent change from baseline
  P-OM3 + simvastatin 80 mg/d | -51.0 [-57.19 to -47.1]
  P-OM3 + simvastatin 20 mg/d | -40.8 [-45.98 to -36.17]
  Placebo + simvastatin 20 mg/d | -34.9 [-40.00 to -30.42]
Statistical Analysis 1: Comparison: Omacor 4 Grams/Day Plus Simvastatin 80 mg/Day; Test type: Superiority — All statistical significance were completed at the 5% level, two-tailed. Comparability of baseline characteristics between those who did and did not opt to enter the extension study was assessed with the chi square test and analysis of variance; p = 0.0008, ANOVA — Threshold for statistical significance p<0.05

2. Secondary Outcome: Median % Change in Non-HDL-C From Baseline to Week 52 by Final Dose of Simvastatin
Description: The median percent change in non-HDL-C from baseline (average of weeks -2, -1, and 0) of the PRV-06009 (NCT00487591) double-blind study to week 52 of PRV-06009X open-label treatment
Time Frame: 52 weeks
Population: Subjects received Omacor 4 grams/day plus simvastatin 80 mg/day for 6 weeks. Simvastatin dose adjusted to 80 mg/day or 40 mg/day at Investigator's discretion after week 6.
  14 participants provided data at Week 6. However, by Week 52, one participant from the 80 mg/day simvastatin group dropped out, leaving a total of 13 participants who completed Week 52.
Measure: Median (95% Confidence Interval); unit: Median percent change from baseline
Groups:
- Omacor 4 Grams/Day Plus Simvastatin 40 mg/Day (Final Dose): Subjects who had successfully completed a 12-wk double-blind crossover study of P-OM3 plus simvastatin 20 mg/d were eligible for the open-label extension study. Omacor 4 grams/day plus simvastatin 80 mg/day. Simvastatin dose adjusted at Investigator discretion after week 6.
  Omacor + 40 mg/day simvastatin: Started with Omacor 4 grams/day plus simvastatin 80 mg/day. Simvastatin dose adjusted at Investigator discretion after week 6. Participants in this arm received an adjusted dose of simvastatin at 40 mg/day for the remainder of the study.
- Omacor 4 Grams/Day Plus Simvastatin 80 mg/Day (Final Dose): Subjects who had successfully completed a 12-wk double-blind crossover study of P-OM3 plus simvastatin 20 mg/d were eligible for the open-label extension study. Omacor 4 grams/day plus simvastatin 80 mg/day. Simvastatin dose adjusted at Investigator discretion after week 6.
  Omacor + 80 mg/day simvastatin: Started with Omacor 4 grams/day plus simvastatin 80 mg/day. Simvastatin dose adjusted at Investigator discretion after week 6. Participants in this arm maintained simvastatin at 80 mg/day for the remainder of the study.
Arm/Group | Omacor 4 Grams/Day Plus Simvastatin 40 mg/Day (Final Dose) | Omacor 4 Grams/Day Plus Simvastatin 80 mg/Day (Final Dose)
Number analyzed (Participants) | 7 | 6
Median percent change from baseline | -50.33 [-58.49 to -43.39] | -40.39 [-53.33 to -36.04]

3. Secondary Outcome: Median % Change in Non-HDL-C From Baseline to Week 104
Description: The median percent change in non-HDL-C from baseline (average of weeks -2, -1, and 0) of the PRV-06009 (NCT00487591) double-blind study to week 104 of PRV-06009X open-label treatment
Time Frame: 104 weeks
Population: Subjects received Omacor 4 grams/day plus simvastatin 80 mg/day for 6 weeks. Simvastatin dose adjusted to 80 mg/day or 40 mg/day at Investigator's discretion after week 6.
  14 participants provided data at Week 6. However, by Week 104, one participant from the 80 mg/day simvastatin group dropped out, leaving a total of 13 participants who completed Week 104.
Measure: Median (95% Confidence Interval); unit: Median percent change from baseline
Groups:
- Omacor 4 Grams/Day Plus Simvastatin 40 mg/Day (Final Dose): Subjects who had successfully completed a 12-wk double-blind crossover study of P-OM3 plus simvastatin 20 mg/d were eligible for the open-label extension study. Omacor 4 grams/day plus simvastatin 80 mg/day. Simvastatin dose adjusted at Investigator discretion after week 6.
  Omacor + simvastatin: Omacor 4 grams/day plus simvastatin 80 mg/day. Simvastatin dose adjusted at Investigator discretion after week 6. Participants in this arm received an adjusted dose of simvastatin at 40 mg/day for the remainder of the study.
- Omacor 4 Grams/Day Plus Simvastatin 80 mg/Day (Final Dose): Subjects who had successfully completed a 12-wk double-blind crossover study of P-OM3 plus simvastatin 20 mg/d were eligible for the open-label extension study. Omacor 4 grams/day plus simvastatin 80 mg/day. Simvastatin dose adjusted at Investigator discretion after week 6.
  Omacor + simvastatin: Omacor 4 grams/day plus simvastatin 80 mg/day. Simvastatin dose adjusted at Investigator discretion after week 6. Participants in this arm maintained simvastatin at 80 mg/day for the remainder of the study.
Arm/Group | Omacor 4 Grams/Day Plus Simvastatin 40 mg/Day (Final Dose) | Omacor 4 Grams/Day Plus Simvastatin 80 mg/Day (Final Dose)
Number analyzed (Participants) | 7 | 6
Median percent change from baseline | -53.46 [-59.45 to -40.17] | -51.25 [-58.93 to -43.56]

ADVERSE EVENTS:
Time Frame: 104 weeks
Description: Subjects reported adverse events at each clinic visit through Week 104
Groups:
- Omacor 4 Grams/Day Plus Simvastatin (40 or 80 mg/Day): Subjects who had successfully completed a 12-wk double-blind crossover study of P-OM3 plus simvastatin 20 mg/d were eligible for the open-label extension study.
  All subjects received Omacor 4 grams/day plus simvastatin 80 mg/day for the first 6 weeks followed by Omacor 4 grams/day plus simvastatin 80 mg/day or Omacor 4 grams/day plus simvastatin 40 mg/day. Assignment to 80 or 40 mg/day simvastatin after Week 6 was based on investigator's assessment of treatment needs.
  The adverse events results reported herein are from the 16 participants who started the extension study. 14 participants completed the first 6 weeks of the extension study and 13 participants completed the extension study in its entirety (up to Week 104). The adverse events were not analyzed by dose (i.e., 40 or 80 mg simvastatin) nor were they analyzed by the number of completers. Unfortunately, we no longer have access to our raw data due to a fire at our facility that destroyed our archived files.
Arm/Group | Omacor 4 Grams/Day Plus Simvastatin (40 or 80 mg/Day)
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 10/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omacor 4 Grams/Day Plus Simvastatin (40 or 80 mg/Day) (N=16)
Viral illness (Infections and infestations) | 1 (1)
Heartburn (Gastrointestinal disorders) | 1 (1)
Sprained ankle (Injury, poisoning and procedural complications) | 1 (1)
Belching (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Bee sting (Injury, poisoning and procedural complications) | 1 (2)
Palpitation (Cardiac disorders) | 1 (1)
Abnormal hepatic function (Hepatobiliary disorders) | 1 (1) — elevated GGT
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) — arm pain
Foot wound (General disorders) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Worsening edema (General disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Torn hamstring (Musculoskeletal and connective tissue disorders) | 1 (1)
Foot infection (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
Potential limitations: 1) small sample size, 2) short duration of each treatment period

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No